CLINICAL TRIAL: NCT06455774
Title: The Effect of Wearable Postural Feedback Devices Added to the Exercise Approach on Neck Pain and Proprioception in Office Workers With Nonspecific Chronic Neck Pain
Brief Title: The Wearable Postural Feedback Devices Combined With Exercise in Office Workers With Chronic Neck Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Selin Uz Tuncay, MSc, PhD Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/06
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain
Keywords: cervical pain; posture; exercise; vibrotactile; feedback
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1- Exercise and Wearable Postural Feedback Devices Group (Experimental): Participants will wear the postural feedback device for 8 weeks, 3 days a week during their desk work (6-8 hours) and will be included in an exercise program including 30 minutes of stretching and strengthening exercises for the cervical region. Exercises will be performed 3 days a week for 30 minutes and will be supervised by a physiotherapist one day a week.
  Interventions: Device: Wearable Postural Feedback Device; Other: Exercise
- Group2- Exercise Group (Experimental): Participants will receive an exercise program consisting of stretching and strengthening exercises for the cervical region. Exercises will be performed 3 days a week for 30 minutes and will be supervised by a physiotherapist one day a week. Patients will be followed up with an exercise diary.
  Interventions: Other: Exercise

INTERVENTIONS:
Device: Wearable Postural Feedback Device — The postural feedback wearable device we will use in the study is programmed to vibrate when hunched postures are detected (based on changes in the curvature and curvature of the spine), alerting users to changes in their body position.
  Arms: Group1- Exercise and Wearable Postural Feedback Devices Group
Other: Exercise — Trapezius, Sternocleidomastoid (SCM), Scalene, pectoral muscles will be targeted for stretching exercises and deep neck flexors, Trapezius, Levator Scapula, Rhomboids will be targeted for strengthening exercises. The intensity of the exercises will be increased according to the weeks. Stretching exercises will be performed as a single set at the pain limit, maintaining the position of the muscle groups in the longest tolerable position for 30 seconds. In strengthening exercises, participants will hold the position for 5-10 seconds at the end of the movement. Moderate resistance elastic bands and free weights will be used for resistance exercises. In the following weeks, progression will be made in all exercises according to the patient's condition.

SUMMARY:
The goal of this clinical trial is to investigate the effects of wearable postural feedback devices added to exercise approach on neck pain and proprioception in office workers with nonspecific chronic neck pain.

H0: The effects of wearable postural feedback devices added to exercise and exercise approach on neck pain and proprioception are similar in office workers with nonspecific chronic neck pain.

H1: The effects of wearable postural feedback devices added to exercise and exercise approach on neck pain and proprioception are different in office workers with nonspecific chronic neck pain.

58 office workers aged 25-55 years with nonspecific chronic neck pain will be included and divided into 2 groups, physiotherapy programs will be applied for 8 weeks, 3 days a week. All participants will be trained on office ergonomics and proper sitting posture at the beginning of the study. Group 1: Exercise and Postural feedback, Group 2: Exercise. Sociodemographic information will be questioned, pain, neck proprioception, craniovertebral angle, neck muscle strength, endurance and range of motion will be assessed. Neck disability index, physical activity level, stress perception level, fatigue level, work performance and patient satisfaction will also be evaluated at baseline and 8 weeks.

DETAILED DESCRIPTION:
Treatment of work-related musculoskeletal disorders can be challenging due to multiple underlying risk factors like physical workload, poor posture, altered sensorimotor control, biopsychosocial conditions. When the information provided by the individual's own sensory system is insufficient, the use of extrinsic feedback has been proposed as an option to reduce sensorimotor discomfort and thus improve movement control. Due to the progress in miniaturization technology of the microelectromechanical system, postural feedback devices have been developed.

Recent studies have used different feedback methods to improve posture. Studies have compared the effectiveness of different types of feedback, active exercise and passive therapy. However, there is a need for studies examining the effects of adding postural feedback to different intervention strategies in the office environment.

Small, lightweight and easy to wear feedback devices can be expected to provide positive effects on neck pain and proprioception in addition to classical exercises by providing real-time feedback to the user during daily activities.

ELIGIBILITY:
Inclusion Criteria:

* Complained of neck pain during work for at least 3 months,
* Neck pain severity of 3 and above according to the Numerical Pain Rating Scale,
* Office worker between the ages of 25-55,
* Full-time and regular desk worker for the last 3 years,
* Participants who use a computer at a desk for at least 3 hours a day will be included.

Exclusion Criteria:

* Having neurological and rheumatologic chronic diseases,
* Receiving physical therapy in the last 6 months
* History of trauma to the upper extremities and spine,
* Having diagnoses such as thoracic outlet, cervical rib, vertebrobasilar artery insufficiency,
* History of cervical spine surgery,
* Having suffered a whiplash injury,
* Diagnosed cervical disc and spine pathologies (such as radiculopathy, myelopathy, fracture, infection, tumor, inflammatory diseases, osteoporosis)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Neck Pain | 8 week
  Neck pain will be assessed using the Numeric Pain Rating Scale. The patient is asked to rate the severity of pain out of 10. The patient chooses the appropriate value between 0; no pain and 10; the worst pain felt. The Neck Pain Numeric Pain Rating Scale has been reported as a valid and reliable method in patients with neck pain.
Proprioception | 8 week
  Neck proprioception will be assessed with the Cervical Joint Position Error Test. Participants will be asked to sit in a chair placed 90 cm from the wall and hold their head in a relaxed neutral position while facing the wall in front of them. A laser pointer will be attached to his/her head with an elastic strap. The laser light on the wall will be marked as the reference point and the participant will then be asked to perform active neck movements (flexion, extension, rotation) and then align the laser light to the reference point with eyes open. He/she will then be asked to repeat the same process with eyes closed and when he/she brings his/her head to the reference point, the new point on the wall will be marked as the target point. The joint position error will be found by measuring the distance between the target and the reference point in cm. Each procedure will be performed 3 times and average values will be taken.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 8 weeks
  Pressure pain threshold will be measured using an algometry device. Pressure pain threshold with algometry is used as a valid and reliable measurement tool for the assessment of pain sensitivity in the neck region. It will be evaluated right and left over the middle part of the upper trapezius muscle (midpoint of the distance between C7 and acromion). Waiting 30 seconds between each measurement taken from the specified area, 3 measurements will be taken and the average value will be recorded.
Craniovertebral Angle | 8 weeks
  Craniovertebral angle will be measured in a standing position using photogrammetry technique. A digital camera will be placed at a distance of 1.5 meters on a stable base, the height of the camera will be adjusted to shoulder level and individuals will be asked to look at a point in front of them to ensure correct posture. A marker will be attached to the C7 spinous process and the targa of the ear of the participants and the craniovertebral angle will be determined from the photographs taken.
Neck Disability Index: | 8 weeks
  Neck Disability Index is a valid and reliable scale used to determine activity limitations due to neck pain. It assesses the level of neck disability in 10 different situations and functions, including pain intensity, self-care, lifting, reading, headache, concentration, work, driving, sleep and leisure activities. Each item is scored from 0 (activity limitation/no disability) to 5 (significant activity limitation/severe disability). The total score ranges from 0-50. In the categorical classification of the total score, 0- 4 indicates no disability, 5-14 indicates mild disability, 15-24 indicates moderate disability, 25-34 indicates severe disability and ≥35 indicates complete disability. A Turkish version and cultural adaptation have been made and its validity and reliability have been demonstrated in individuals with neck pain.
Muscle strength | 8 weeks
  Maximal isometric muscle strength of cervical region flexor and extensor muscles will be measured with a hand-held dynamometer. Cervical flexor muscle strength will be measured with the participants in supine position, head and neck in neutral position, knee flexion and arms at the side of the body. Cervical extensor muscle strength will be measured with the participants in the prone position with arms at the side of the body. During the measurements, participants will be asked to generate maximum force against the dynamometer device throughout the test (3-5 seconds). In flexor and extensor muscle strength measurements, three measurements will be made with a one-minute rest period between each measurement and their averages will be recorded. It has been reported that measuring maximal isometric muscle forces of flexor and extensor muscles in the cervical region with a hand-held dynamometer is a reliable and easy-to-apply method.
Range of motion | 8 weeks
  Normal range of motion of the cervical joints was measured using a 360-degree universal goniometer. Normal range of motion of the cervical joints will be measured in the flexion, extension, rotation and lateral flexion directions with the participants in a sitting position, head and trunk held upright.
Physical activity level | 8 weeks
  The physical activity levels of the participants will be assessed using the 'International Physical Activity Index short form' whose validity and reliability studies were conducted by Craig et al. In this questionnaire, the time spent in sitting, walking, moderately vigorous and vigorous activities during the last seven days is questioned. Turkish validity and reliability of the questionnaire was performed.
Stress Perception Level | 8 weeks
  The stress perception level of the participants will be assessed with the 'Perceived Stress Scale'. The questionnaire, which consists of 14 items in total, evaluates the level of stress perception in certain situations in one's life. Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". Survey scores range from 0 to 56. A high score indicates a high level of stress perception (Cohen et al., 1983). Turkish validity and reliability study of the questionnaire was conducted (Eskin et al., 2013).
Fatigue Assessment | 8 weeks
  The fatigue level of the participants will be assessed using the 'Fatigue multidimensional assessment scale' (Piper et al., 1989). Turkish validity and reliability study of the scale in chronic musculoskeletal diseases has been conducted (Yildirim & Ergin, 2013).
Work performance | 8 weeks
  Participants' work performance will be assessed with the Health and Work Performance Scale. The short version of the scale developed by the World Health Organization consists of 11 items answered in two different types. The scale assesses employees' work productivity with two subscales (Kessler et al., 2003). The absenteeism part consists of 8 items and measures the time spent on work and lost time as numerical values. The absenteeism part consists of 3 items and evaluates the quality of the work done during the work process. This section is measured by scoring between 0 (worst) and 10 (best). In the scale, the evaluation process can be done for a seven-day period and for a four-week period. The scale has been shown to be valid and reliable for white-collar employees in Turkey (Kuru, 2019).
Patient Satisfaction | 8 week
  The level of satisfaction of all study participants with the treatment they received at the end of the study will be assessed with the Global Change Scale. It is a scale in which patients determine the amount of improvement or deterioration in their health status over time from their own perspectives. Global change scales are widely used in clinical research, especially in the musculoskeletal system. There are different rating scales. In this study, an 11-unit scale will be used (-5: much worse, 0: same, +5: completely improved).

CONTACTS AND LOCATIONS:
Overall Officials: Gökşen Kuran Aslan, Prof, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No